CLINICAL TRIAL: NCT00385190
Title: An Ascending Multiple Dose Study of the Safety, Tolerability, and Pharmacokinetics of Study Drug Administred Orally to Healthy Japanese Male Subjects
Brief Title: Study Evaluating the Pharmacokinetics of HCV-796 in Healthy Japanese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3173A1-108
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: SAD
MeSH Terms: interventions — HCV 796

INTERVENTIONS:
Drug: HCV-796

SUMMARY:
The purpose of the study is to assess the safety and tolerability of ascending multiple oral doses of HCV-796 in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead ECG.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2006-07; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Safety and pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Minato-ku, Tokyo, Japan